CLINICAL TRIAL: NCT00417144
Title: Randomized Controlled Trial Comparing the Effect of GnRH Agonist and Antagonist Ovarian Stimulation Protocols in PCOS Patients
Brief Title: Comparison Between GnRH Agonist and GnRH Antagonist Protocols of Ovarian Stimulation in PCOS Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eugonia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ag vs antag PCOS
Record Dates: First submitted 2006-12-22; First posted 2006-12-29 (Estimated); Last update posted 2006-12-29 (Estimated); Status verified 2006-12

CONDITIONS: Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome
Keywords: OHSS; PCOS; GnRH antagonist; GnRH agonist
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome | interventions — Triptorelin Pamoate; ganirelix

INTERVENTIONS:
Drug: Arvekap 0.1mg (Triptorelin, Ipsen, France)
Drug: Ganirelix 0.25mg (Orgalutran, Organon, The Netherlands)

SUMMARY:
The purpose of this study is to compare pregnancy rates and the occurrence of OHSS in PCOS patients who were treated with GnRH agonist and GnRH antagonist protocols ovarian stimulation during an IVF cycle. Our hypothesis is that the GnRH antagonist protocol reduces the occurrence and severity of OHSS compared to the GnRH agonist protocol.

DETAILED DESCRIPTION:
Women with polycystic ovarian syndrome (PCOS) represent a group of patients at high risk of developing ovarian hyperstimulation syndrome (OHSS), an iatrogenic complication of ovarian stimulation during IVF treatment. In contrast to mild OHSS, severe OHSS is a life-threatening complication, characterized by massive ovarian enlargement, ascites, pleural effusion, oliguria, haemoconcentration and thromboembolic phenomena. Currently, no curative therapy for OHSS is available and thus prevention is considered the most effective "treatment". Several measures have been adopted to reduce the occurrence of the syndrome, the most effective being cycle cancellation and withholding of human chorionic gonadotropin (hCG), which seems to be the most critical factor for the development of OHSS.

COMPARISON: This study aims to compare the development and severity of OHSS, as well as ongoing pregnancy rates in PCOS patients who received a flexible GnRH antagonist (Ganirelix) protocol vs a long GnRH agonist (Arvekap) protocol of ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PCOS (presence of oligo-ovulation/anovulation and polycystic ovaries)

Exclusion Criteria:

* Normal responders
* Poor responders

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200
Dates: Start 2003-11; Study Completion 2007-05

PRIMARY OUTCOMES:
Development of OHSS
Ongoing pregnancy rate per embryo transfer

SECONDARY OUTCOMES:
Biochemical pregnancy
Clinical pregnancy
Embryological data

CONTACTS AND LOCATIONS:
Overall Officials: Tryfon Lainas, PhD, Principal Investigator — Eugonia
Locations (1):
- Eugonia, Athens, Greece

REFERENCES:
- [Background] Aboulghar MA, Mansour RT. Ovarian hyperstimulation syndrome: classifications and critical analysis of preventive measures. Hum Reprod Update. 2003 May-Jun;9(3):275-89. doi: 10.1093/humupd/dmg018. PMID 12859048
- [Derived] Lainas TG, Sfontouris IA, Zorzovilis IZ, Petsas GK, Lainas GT, Alexopoulou E, Kolibianakis EM. Flexible GnRH antagonist protocol versus GnRH agonist long protocol in patients with polycystic ovary syndrome treated for IVF: a prospective randomised controlled trial (RCT). Hum Reprod. 2010 Mar;25(3):683-9. doi: 10.1093/humrep/dep436. Epub 2009 Dec 15. PMID 20008886